CLINICAL TRIAL: NCT07230600
Title: Autologous Adipose-derived Stromal Vascular Fraction Therapy for Refractory Endometrial Infertility
Brief Title: AD-SVF Therapy for Refractory Endometrial Infertility
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yali Hu, M.D., Ph.D., The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC2025-006-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Endometrium; Atrophy; Intrauterine Synechiae
Keywords: adipose-derived stromal vascular fraction; thin endometrium
MeSH Terms: conditions — Atrophy; Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AD-SVF therapy (Experimental): AD-SVF intrauterine infusion therapy
  Interventions: Biological: AD-SVF

INTERVENTIONS:
Biological: AD-SVF — AD-SVF is isolated and extracted from adipose tissue for intrauterine infusion therapy.

SUMMARY:
The purpose of this study is to initially explore the efficacy of adipose-derived stromal vascular fraction (AD-SVF) therapy in the treatment of refractory endometrial infertility.

DETAILED DESCRIPTION:
Patients with refractory thin endometrium (endometrial thickness < 6 mm at late proliferative phase or after high-dose estrogen therapy) and/or moderate to severe intrauterine adhesion are recruited for fertility. After detailed explanation of the treatment plan, written informed consent will be obtained from the patients. The subjects undergo liposuction performed by plastic surgeons to obtain adipose tissue, from which AD-SVF is isolated and extracted for intrauterine infusion therapy. Six months post-AD-SVF treatment, the improvement in menstrual volume and endometrial thickness will be assessed during follow-up visits. The subjects will be advised, based on their personal inclination, to attempt conception (hysteroscopic surgery will be repeated if necessary), and their early pregnancy outcomes will be documented in subsequent follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. refractory thin endometrium (endometrial thickness < 6 mm on the day of ovulation or the day of endometrial transformation during a hormone replacement cycle) and/or moderate to severe intrauterine adhesion；
2. Inability to undergo autologous bone marrow stem cells-scaffold (BMSC) transplantation due to failed bone marrow aspiration, or lack of significant effect following the BMSC treatment;
3. with fertility intentions;
4. normal ovarian function or availability of cryopreserved embryos;
5. 18kg/m^2 < body mass index (BMI) < 30kg/m^2;

Exclusion Criteria:

1. Chromosomal karyotype abnormalities in one spouse;
2. Severe endometriosis, uterine fibroids affecting the uterine cavity morphology, or uterine malformations;
3. Abnormalities in coagulation function, hepatic or renal function, or other underlying conditions deemed by the investigator to potentially impact the study's progression (uncontrolled hypertension, diabetes, autoimmune diseases, etc.);
4. Contraindications for pregnancy;
5. Contraindications for hormonal cycle therapy;
6. History of pelvic tumors;
7. Simultaneous participation in other clinical studies.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with endometrial thickness of 6 mm or greater | 6 months after AD-SVF intrauterine infusion therapy
  During the late proliferative phase, the endometrial thickness between anterior and posterior uterine walls is measured to be at least 6 mm through a median sagittal section of the uterus at least once.

SECONDARY OUTCOMES:
Menstrual flow score at the 2nd month post-treatment | 2 months after AD-SVF intrauterine infusion therapy
  2 months after treatment, menstrual flow is scored according to the Pictorial Blood-loss Assessment Chart, with scores ranging from 0 to 100, and higher scores indicate better outcomes.
Menstrual flow score at the 6th month post-treatment | 6 months after AD-SVF intrauterine infusion therapy
  6 months after treatment, menstrual flow is scored according to the Pictorial Blood-loss Assessment Chart, with scores ranging from 0 to 100, and higher scores indicate better outcomes.
Chemical pregnancy | 9 months after AD-SVF intrauterine infusion therapy
  Serum β-HCG ≥ 10 mIU/mL is detected at least 30 days after menstruation.
Clinical pregnancy | 9 months after AD-SVF intrauterine infusion therapy
  Ultrasound indicates the presence of a gestational sac and fetal heartbeat in the uterine cavity Ultrasound indicates the presence of a gestational sac and fetal heartbeat in the uterine cavity Ultrasound indicates the presence of a gestational sac and fetal heartbeat in the uterine cavity at 6-8 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University; Huiyan Wang, Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China